CLINICAL TRIAL: NCT03400241
Title: Pharmacokinetic Pilot Study Comparing Absorption of Inhaled Tiotropium Between Tiotropium Easyhaler® Products and Spiriva® Capsules Delivered Via HandiHaler®
Brief Title: Pharmacokinetic Study Comparing Tiotropium Easyhaler and Spiriva Handihaler
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Orion Corporation, Orion Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 3122002
Record Dates: First submitted 2018-01-09; First posted 2018-01-17 (Actual); Last update posted 2018-06-14 (Actual); Status verified 2018-06

CONDITIONS: Healthy Subjects

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Tiotropium Easyhaler Product A (Experimental): tiotropium bromide monohydrate 2 inhalations as a single dose
  Interventions: Drug: Tiotropium Bromide Monohydrate
- Tiotropium Easyhaler Product B (Experimental): tiotropium bromide monohydrate 2 inhalations as a single dose
  Interventions: Drug: Tiotropium Bromide Monohydrate
- Tiotropium Easyhaler Product C (Experimental): tiotropium bromide monohydrate 2 inhalations as a single dose
  Interventions: Drug: Tiotropium Bromide Monohydrate
- Spiriva HandiHaler (Active Comparator): tiotropium bromide monohydrate 2 Spiriva capsules inhaled via HandiHaler
  Interventions: Drug: Tiotropium Bromide Monohydrate

INTERVENTIONS:
Drug: Tiotropium Bromide Monohydrate — Tiotropium Easyhaler 10 mcg/dose Product A
  Arms: Tiotropium Easyhaler Product A
Drug: Tiotropium Bromide Monohydrate — Tiotropium Easyhaler 10 mcg/dose Product B
  Arms: Tiotropium Easyhaler Product B
Drug: Tiotropium Bromide Monohydrate — Tiotropium Easyhaler 10 mcg/dose Product C
  Arms: Tiotropium Easyhaler Product C
Drug: Tiotropium Bromide Monohydrate — Spiriva 18 Mcg/capsule inhaled via HandiHaler
  Arms: Spiriva HandiHaler

SUMMARY:
Absorption of inhaled tiotropium is compared between three Tiotropium Easyhaler products and Spiriva capsules inhaled via HandiHaler. All subjects will receive all products as a single dose.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female subjects
* 18-60 years old
* Body mass index >19 and <30 kg/m2
* Weight at least 50 kg
* Written informed consent obtained

Exclusion Criteria:

* Evidence of a clinically significant cardiovascular, renal, hepatic, haematological, gastrointestinal, pulmonary, metabolic, endocrine, neurological or psychiatric disease.
* Any condition requiring regular concomitant treatment.
* Any clinically significant abnormal laboratory value or physical finding that in the opinion of the investigator may interfere with the interpretation of study results or constitute a health risk for the subject.
* Known hypersensitivity to tiotropium bromide, atropine or its derivatives, or lactose.
* Pregnant or lactating females and females of childbearing potential not using proper contraception.
* Blood donation, loss of a significant amount of blood or administration of another investigational medicinal product within 90 days before the first study treatment administration

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2018-02-19 (Actual); Primary Completion 2018-04-18 (Actual); Study Completion 2018-04-18 (Actual)

PRIMARY OUTCOMES:
Peak plasma concentration (Cmax) of tiotropium | between 0-72 hours after dosing
Area under the concentration-time curve (AUC) of tiotropium from time zero to 72 h after the study treatment administration | 0-72 hours after dosing
Truncated area under the concentration-time curve (AUC) of tiotropium from time zero to 30 min after study treatment administration | 0-30 minutes after dosing

SECONDARY OUTCOMES:
Time to reach peak concentration in plasma (tmax) of tiotropium | between 0-72 hours after dosing

OTHER OUTCOMES:
Adverse events | throughout the study, an average of 10 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ulla Sairanen, MSc, Study Director — Orion Corporation, Orion Pharma
Locations (1):
- Clinical Pharmacology Unit, Espoo, Finland